CLINICAL TRIAL: NCT04493151
Title: Pharmacokinetics of Imipenem/Cilastatin/Relebactam in Critically Ill Patients Receiving Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Imipenem/Cilastatin/Relebactam PK in ECMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph L. Kuti, PharmD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Joseph L. Kuti, PharmD, Associate Director, Center for Anti-Infective Research and Development, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 59752
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: beta-lactam; pharmacokinetics
MeSH Terms: conditions — Sepsis | interventions — imipenem, cilastatin and relebactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imipenem-Cilastatin-Relebactam (Experimental): Participants will receive a four to six doses of intravenous imipenem-cilastatin-relebactam as per current prescribing information based on estimated creatinine clearance.
  Interventions: Drug: Imipenem, Cilastatin and Relebactam

INTERVENTIONS:
Drug: Imipenem, Cilastatin and Relebactam — After receipt of imipenem-cilastatin-relebactam, ten blood samples will be collected to determine the pharmacokinetics of imipenem and relebactam.
  Other Names: Recarbrio

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a from of cardiopulmonary life-support for critically ill patients where blood is extracted from the vascular system and circulated by a mechanical pump while it is oxygenated and re-infused into the patient's circulation. It is well known that critically ill patients may experience alterations in antibiotic pharmacokinetics, and as a result, dosing modifications are generally required. There is a need to understand how ECMO circuits affect the pharmacokinetics and disposition of drugs. This study is designed to assess the pharmacokinetics of the new broad-spectrum antibiotic, imipenem-cilastatin-relebactam, in critically ill patients receiving ECMO.

DETAILED DESCRIPTION:
This is a single center, open-label study to determine imipenem-cilastatin-relebactam pharmacokinetics in critically ill patients receiving ECMO. Eight patients with suspected suspected sepsis and who are receiving ECMO will be enrolled. Each participant will receive four to six doses of imipenem-cilastatin-relebactam according to current approved prescribing information, followed by ten blood samples to determine concentrations. Non-compartmental and population pharmacokinetic analyses will be determined to assess the effects of ECMO on imipenem and relebactam pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* On support with Veno-venous- or Veno-arterial-ECMO;
* Documented infection or presumed infection as confirmed by the presence of at least one of the following criteria within the past 72 hours:

  * Documented fever (oral, rectal, tympanic, or core temperature > 38.5° C)
  * Hypothermia (oral, rectal, tympanic, or core temperature < 35.0° C)
  * An elevated white blood cell (WBC) count ≥ 12,000 cells/mm3

Exclusion Criteria:

* If female, currently pregnant or breast feeding;
* History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam agent (a history of mild rash to a β-lactam followed by uneventful re-exposure is not a contraindication);
* Severe renal dysfunction defined as a creatinine clearance < 15 mL/min (calculated by the Cockcroft-Gault equation using actual body weight) or requirement for continuous renal replacement therapy or hemodialysis;
* Hemoglobin less than 8 mg/dL at baseline;
* Use of probenecid, valproic acid, or imipenem within 3 days before study drug infusion;
* Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal;
* Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator);
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data;
* Planned or prior participation in any other interventional drug study within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imipenem-Cilastatin-Relebactam
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imipenem-Cilastatin-Relebactam
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Imipenem Clearance
Description: The clearance in liters/hour of imipenem from the plasma of critically ill patients receiving ECMO.
Time Frame: 6 hours (samples collected before the first imipenem/cilastatin/relebactam dose (i.e., blank), and at 0.5 and 6 hours following the first dose, and then at 0, 0.5, 0.75, 1, 2, 4, 5, and 6 hours after the start of the final dose).
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Imipenem-Cilastatin-Relebactam
Number analyzed (Participants) | 7
Liters per hour | 15.21 (6.52)

2. Primary Outcome: Relebactam Clearance
Description: The clearance in liters/hour of relebactam from the plasma of critically ill patients receiving ECMO.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Imipenem-Cilastatin-Relebactam
Number analyzed (Participants) | 7
Liters per hour | 6.95 (1.34)

3. Secondary Outcome: Imipenem Area Under the Curve (AUC)
Description: The AUC in milligram*hour/liter of imipenem calculated from concentrations collected between zero and 6 hours at steady-state
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Imipenem-Cilastatin-Relebactam
Number analyzed (Participants) | 7
mg*h/L | 36.9 (13.3)

4. Secondary Outcome: Relebactam Area Under the Curve (AUC)
Description: The AUC in milligram*hour/liter of relebactam calculated from concentrations collected between zero and 6 hours at steady-state
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Imipenem-Cilastatin-Relebactam
Number analyzed (Participants) | 7
mg*h/L | 45.3 (33.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 48 hour window, from the first imipenem-relebactam dose (0 hour) to the end of blood sampling (6 hours), plus an 24 hour observation window after the last sample was collected, culminating with physical exam. Note: 8 subjects were enrolled and received imipenem-relebactam. Although only 7 subjects were included in results analysis due to inability to obtain blood samples in 1 subject, all 8 subjects are included in the adverse event reporting.
Description: Adverse event - any pathologic or unintended change in the structure (signs), function (symptoms), or chemistry (laboratory values) of the body associated with the use of the study drug, whether or not considered drug related: MILD - present, but easily tolerated MODERATE - discomfort that interferes with usual activities SEVERE - incapacitating, inability to work or do usual activities
Arm/Group | Imipenem-Cilastatin-Relebactam
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imipenem-Cilastatin-Relebactam (N=8)
Alkaline Phosphate Increase (Hepatobiliary disorders) | 1 (1)
C. difficile Diarrhea (Gastrointestinal disorders) | 1 (1)
Increasing Leukocytosis (Infections and infestations) | 2
Aspartate Aminotransferase Increase (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A study limitation is the protocol defined exclusion of patients on concomitant continuous renal replacement therapy (CRRT), which is common in patients receiving ECMO (extracorporeal membrane oxygenation). Dosing modifications may be necessary in patients receiving both CRRT and ECMO.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT04493151/Prot_SAP_000.pdf